CLINICAL TRIAL: NCT03819686
Title: Reducing Disparities in Living Donor Transplant Among African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kimberly R Jacob Arriola, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00098952; R01DK114891 (NIH)
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant
Keywords: end stage renal disease; ESRD; living donor kidney transplantation; LDKT; African American
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Living ACTS website (Experimental): In addition to the provision of standard transplant education procedures, a patient will watch the Living ACTS video (embedded in the Living ACTS website) along with any family members or friends who are accompanying a patient. Plus minimum of 5 minutes navigating the website (aside from watching the 20-minute video).
  Interventions: Behavioral: Living ACTS website; Behavioral: Standard transplant education procedures
- Standard transplant education procedures (Other): Usual Care, which involves the provision of standard transplant education procedures at each transplant center, which entail reviewing a packet of information with the pre-transplant coordinator. The packet serves to inform transplant candidates and their families about the option living donor kidney transplantation (LDKT). In addition, participants will be provided an iPad/tablet to watch two 10-minute National Kidney Foundation videos about kidney disease and transplantation in their private room during their regularly scheduled KT evaluation. This video discusses information about transplant, but does not specifically address LDKT and is not culturally-sensitive to African American population.
  Interventions: Behavioral: Standard transplant education procedures

INTERVENTIONS:
Behavioral: Living ACTS website — Living ACTS: About Choices in Transplantation and Sharing video that draws from the Information-Motivation-Behavioral Skills Model of individual level behavior change. A patient will watch the Living ACTS video (embedded in the Living ACTS website) along with any family members or friends who are accompanying a patient. Plus minimum of 5 minutes navigating the website (aside from watching ~20-minutes of videos from the website)
  Arms: Living ACTS website
Behavioral: Standard transplant education procedures — Review of a packet of information with the pre-transplant coordinator. The packet serves to inform transplant candidates and their families about the option living donor kidney transplantation (LDKT). In addition, participants will be provided an iPad/tablet to watch two ~10-minute National Kidney Foundation videos about kidney disease and transplantation in their private room during their regularly scheduled KT evaluation. This video discusses information about transplant, but does not specifically address LDKT and is not culturally-sensitive to African American population.

SUMMARY:
For most of the patients in the United States with end stage renal disease (ESRD), kidney transplantation represents the optimal treatment, and living donor kidney transplantation (LDKT) is preferable. Nevertheless, there are pervasive racial disparities in access to LDKT. The main outcome of this study is change in the proportion of study participants who have at least one living donor inquiry by friends/family over study period.The long-term objective is to understand the combined effect of a systems-level intervention (Transplant Referral EXchange or T-REX) and a culturally-sensitive individual-level educational intervention (web-based Living ACTS: About Choices in Transplantation and Sharing) on racial disparities in access to LDKT.

DETAILED DESCRIPTION:
For most of the patients in the United States with end stage renal disease (ESRD), kidney transplantation represents the optimal treatment. Moreover, living donor kidney transplantation (LDKT) offers numerous advantages such as better kidney quality, increased short- and long-term graft survival, lower rates of acute rejection, and reduced health care cost. Nevertheless, there are pervasive racial disparities in access to LDKT, with white ESRD patients four times more likely to receive a LDKT than African American ESRD patients. The main outcome of this study is change in the proportion of study participants who have at least one living donor inquiry by friends/family over 12 months from baseline.The long-term objective is to understand the combined effect of a systems-level intervention that enhances communication between dialysis facility and transplant center clinicians (Transplant Referral EXchange or T-REX) and a culturally-sensitive individual-level educational intervention (web-based Living ACTS: About Choices in Transplantation and Sharing) on racial disparities in access to LDKT.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred (from dialysis facility, chronic kidney disease clinic, or self) and scheduled for an evaluation at one of the four study sites within the study time period.
* African American or Black
* age 18 to 70 years
* BMI < 39
* English-speaking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Jacob Arriola, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory Transplant Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arriola KJ, Barrett D, Pastan S, Perryman J, DuBay D, Tresslar C, De Abreu SU, Di M, Teunis L, Montoya M, Mangurenje T, Patzer RE. Immediate Postintervention Outcomes from a Randomized Trial that Sought to Enhance Access to Live Donor Kidney Transplant for Black and African Americans. Prog Transplant. 2025 Mar;35(1):5-12. doi: 10.1177/15269248241304794. Epub 2024 Dec 19. PMID 39698959

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Living ACTS Website | Standard Transplant Education Procedures
Started | 224 | 192
Completed | 222 | 189
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Living ACTS Website | Standard Transplant Education Procedures | Total
Number analyzed (Participants) | 224 | 192 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.83 (11.64) | 49.09 (12.18) | 49.49 (11.88)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 93 | 89 | 182
  Male | 128 | 102 | 230
  Prefer not to answer | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 223 | 192 | 415
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 224 | 192 | 416
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 224 | 192 | 416

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With at Least One Inquiry From a Potential Living Donor
Description: Data collection form that captures potential recipient ID (i.e. study participant), date of living donor inquiry, and donor inquiry ID, will be securely obtained from each transplant center following a 12 month period from enrollment. Data will be collected electronically for all study participants through a secure, HIPAA-compliant data server (QualityNet). The percent of patients with at least one inquiry from a potential living donor among patients who receive Living ACTS will be compared to those who receive a control website with embedded educational video.
Time Frame: Baseline, 12 months
Population: Number of participants analyzed included patients that completed the visit for each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Living ACTS Website | Standard Transplant Education Procedures
Number analyzed (Participants) | 224 | 192
percentage of participants
  Baseline | 15.63 | 15.63
  12 months post-intervention: number analyzed (Participants) | 222 | 189
  12 months post-intervention | 15.77 | 15.87

2. Secondary Outcome: Knowledge and Understanding of Donation/Transplantation Assessment Score
Description: Scale includes 13 true/False questions, score ranges from 0 to 13, 0 Min-13 Maximum where higher scores indicate greater knowledge (i.e., participants receive 1 point for each correct answer).
Time Frame: Baseline, Day 1 immediately post-intervention
Population: Number of participants analyzed included patients that completed the visit for each time point for the purpose of collecting data for this study outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Living ACTS Website | Standard Transplant Education Procedures
Number analyzed (Participants) | 224 | 192
score on a scale
  Knowledge assessment score at baseline | 10.00 (1.49) | 10.18 (1.60)
  Knowledge assessment score at average 12 months post-intervention: number analyzed (Participants) | 222 | 189
  Knowledge assessment score at average 12 months post-intervention | 10.14 (1.45) | 10.03 (1.72)

3. Secondary Outcome: Motivation Scale Score to Ask a Family Member to be a Living Donor
Description: 9-item scale assesses motivation to ask a family member to be a living donor. Potential responses range from 1 to 5, Possible score range from 9 to 45 with higher values indicating stronger agreement with the statement.
Time Frame: Baseline, Day 1 immediately post-intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Living ACTS Website | Standard Transplant Education Procedures
Number analyzed (Participants) | 224 | 192
score on a scale
  Motivation scale score at baseline | 36.03 (5.00) | 35.58 (4.86)
  Motivation scale score at average 12 months post-intervention: number analyzed (Participants) | 222 | 189
  Motivation scale score at average 12 months post-intervention | 37.00 (4.93) | 36.38 (4.98)

4. Secondary Outcome: Confidence in Initiating a Conversation About LDKT
Description: 10-item behavioral skills scale measures confidence in initiating a conversation about LDKT. Potential responses range from 1 to 5, total possible score range is 10-50, with higher values indicate stronger confidence.
Time Frame: Baseline, Day 1 immediately post-intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Living ACTS Website | Standard Transplant Education Procedures
Number analyzed (Participants) | 224 | 192
score on a scale
  Behavioral skills scale score at baseline | 40.38 (7.35) | 39.45 (6.63)
  Behavioral skills scale score at average 12 months post-baseline: number analyzed (Participants) | 222 | 189
  Behavioral skills scale score at average 12 months post-baseline | 41.98 (6.88) | 40.46 (6.85)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Month 12.
Arm/Group | Living ACTS Website | Standard Transplant Education Procedures
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/192
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/192
Other Adverse Events (participants affected / at risk) | 0/224 | 0/192

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT03819686/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT03819686/ICF_000.pdf